CLINICAL TRIAL: NCT06779669
Title: Use of Alternative and Complementary Medicine by Colorectal Cancer Patients
Acronym: ALTERNATIVCCR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI24_0033 (ALTERNATIVCCR)
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Complementary and alternative medicine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Complementary and alternative medicine user (Other): Selected patients will answer a questionnaire about their practice and habits with regard to alternative and complementary medicines. Of these patients, 12 will also complete an additional qualitative questionnaire.
  Interventions: Other: Questionnaire CAM

INTERVENTIONS:
Other: Questionnaire CAM — Selected patients will answer a questionnaire about their practice and habits with regard to alternative and complementary medicines. Of these patients, 12 will also complete an additional qualitative questionnaire.

SUMMARY:
Complementary and alternative medicine (CAM) is defined by the National Center for Complementary and Alternative Medicine as "a group of diverse medical and health systems, practices and products that are not currently considered part of conventional medicine" (Complementary, Alternative, or Integrative Health, n. d. 2012). Complementary medicine is used to complement conventional medicine, and alternative medicine is used instead of conventional medicine (Dy et al., 2004). These are two very different approaches, whose consequences for a cancer patient can be completely different. The use of CAM is steadily increasing in most countries. A study carried out in France in 2017 revealed that for half of CAM users, the diagnosis of cancer was one of the main factors that led patients to turn to CAM (Sarradon-Eck et al., 2017). CAM use was found to be significantly associated with younger age, female gender and higher education (Sarradon-Eck et al., 2017). The source of information about MAC was mainly friends/family and the media, while doctors and nurses played a succinct role in MAC information (Molassiotis et al., 2005). The most frequently cited reasons for using CAM were to improve their physical well-being, strengthen their bodies, improve their emotional well-being and relieve the side effects of treatment (Sarradon-Eck et al., 2020). Another study carried out in 2019 at nine centers in France showed that 45% of glioma patients had changed their eating habits after glioma diagnosis, 44% were on complementary treatment, mainly vitamins and dietary supplements, and 32% were using alternative medicine, mainly magnetism and acupuncture. A total of 68% reported using at least one of these approaches (Le Rhun et al., 2019). Another single-center study conducted in France in 2019 found that 83% of cancer patients used CAM (M et al., 2019). CAM included osteopathy, homeopathy, acupuncture, therapeutic touch, magnetism, naturopathy, cupping, Chinese medicine, reflexology and hypnosis. However, no studies have been carried out to assess the use of CAM among colorectal cancer (CRC) patients in France.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed with colorectal cancer
* To be operated on between 2017 and 2022

Exclusion Criteria:

* The patient refuses to give consent to participate in the study
* Non-primary colorectal cancer (metastasis to the colon or rectum from another primary cancer; cancer originating in the appendix)
* Primary metastatic cancer other than colorectal cancer
* Discovery of cancer synchronous with colorectal cancer
* Guardianship or trusteeship
* Cognitive disorders (Alzheimer's, dementia, etc.)
* Severe psychiatric disorder (neurodevelopmental disorder, psychotic disorder, mood disorder, etc.) according to the specific DSM-5 and ICD-11 classifications
* Severe deafness (unable to answer questions during telephone interview)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
MAC using | Month 2
  Proportion of patients treated at Limoges University Hospital for colorectal cancer (CRC) using MACs

SECONDARY OUTCOMES:
Demographic factors | Month 2
  Demographic factors associated with MAC use (Odds ratio)
Clinical factors | month 2
  Clinical factors associated with MAC use (Odds ratio)
Recurrence time | Month 2
  3-year recurrence time for patients undergoing CRC surgery at Limoges University Hospital (Hazard ratio)
Quality of life | Month 2
  Quality of life assessed by QLQ C30 questionnaire (Odds ratio)
MAC information sources | month 2
  Description of MAC information sources (frequencies and percentages)
Reasons of using MAC | month 2
  Description of the reasons why patients use or do not use these practices (frequencies and percentages)
Effects perceived | month 2
  Description of effects perceived by MAC users (frequencies and percentages)
healthcare professionals' report on MAC | month 2
  Description of healthcare professionals' report on MAC use (frequencies and percentages)

CONTACTS AND LOCATIONS:
Overall Officials: Niki CHRISTOU, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No